CLINICAL TRIAL: NCT03344081
Title: Evaluating Multivariate MRI Maps of Body Awareness: A Pilot Functional Magnetic Resonance Imaging (fMRI) Study of Breath Meditation
Brief Title: Evaluating Multivariate MRI Maps of Body Awareness
Acronym: EMBODY
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Other Study IDs: 15-16716; K08AT009385 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-11-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Attention
Keywords: attention; interoception; meditation; mind wandering

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meditators: Meditators will have practiced meditation for at least the 5 years, at least 90 minutes weekly. They will have completed at least 14 days of retreat practice in the past 5 years. At least half of their meditation practice will include attention to the breath and body. All participants will be MRI-compatible, healthy with no health conditions that affect breathing, have no current psychiatric disorder, and not be taking psychotropic medications.
- Controls: Control participants will be age- and gender-matched to each meditators. They will have little to no previous meditation experience. All participants will be MRI-compatible, healthy with no health conditions that affect breathing, have no current psychiatric disorder, and not be taking psychotropic medications.

SUMMARY:
Meditation skills, or paying attention to internal mental states, are thought to improve people's health. This study is developing a new brain measure of meditation skills, called the EMBODY Task, using functional magnetic resonance imaging (fMRI). The investigators are testing whether pattern recognition methods can be applied to fMRI data to identify mental states during meditation, including attention to the body and to thoughts. This task is being developed in meditation practitioners and non-meditators. The goal is to understand what people are paying attention to during meditation using brain data. The investigators hypothesize that pattern recognition technology will be able to identify different mental states that occur during meditation.

DETAILED DESCRIPTION:
The investigators are developing a new functional magnetic resonance imaging (fMRI) task (the EMBODY Task) to measure mental states during meditation using pattern recognition or machine learning technology. This task is being piloted and validated in 20 meditators and 20 control participants, in two waves of pilot testing. Meditators will have practiced meditation for at least the 5 years, at least 90 minutes weekly. Control participants will have little to no meditation experience and will be age- and gender-matched to each meditator. All participants will be MRI-compatible, healthy with no health conditions that affect breathing, have no current psychiatric disorder, and not be taking psychotropic medications.

In the EMBODY Task, participants will be instructed to pay attention to areas of the body, their thoughts, sounds in the scanner, and to stop paying attention, in short intervals (16-45s). They will also meditate on their breath for 10 minutes. The investigators will determine whether pattern recognition technology can distinguish 5 mental states, and whether these brain patterns can be used to identify mental states during meditation. The investigators hypothesize that all 5 mental states will be distinguished by pattern recognition in the meditators, and potentially in the controls. Investigators also hypothesize that meditators should pay attention to their breath longer during meditation compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, 25-65 years of age.
* Meditators will be affiliated with meditation centers that are based in the Vipassana tradition or Zen traditions. In the past 5 years, meditators will have a consistent practice in mindfulness of body practices, where consistent practice is defined as practicing for at least 90 minutes in a typical week. They will also have had at least 14 days of total silent retreat practice in the past 5 years. At least half of total practice time as reported by the participants will be engaged in mindfulness of body practices (e.g., breath meditation, body scan, mindfulness of emotions, mindful yoga, walking meditation).
* Non-meditator control group. Within the past 3 years, participants will not have engaged in regular meditation (including from courses such as Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, and Dialectical Behavioral Therapy), yoga, or other mind-body practice (such as Tai Chi, Feldenkrais, sensory awareness, or related practices), defined as more than 20 minutes of practice at least two times per week. If there is experience with mind-body practices prior to the past 3 years, it should not include an extended period of consistent practice (such as 20 min daily practice for a year or more) or a period of intensive practice longer than 7 days (e.g., 10-day silent retreat).

Exclusion Criteria:

Participants who endorse:

1. being smokers;
2. chronic or recurrent bronchial or pulmonary disease requiring medical attention;
3. having been diagnosed with sleep apnea;
4. a history of an upper or lower respiratory tract infection in the 6 weeks preceding the study;
5. pregnancy;
6. diseases that restrain chest or abdominal breathing, such as ankylosing spondylitis, systemic lupus, chronic abdominal pain, chronic liver or kidney diseases,
7. can not fit comfortably in the MRI scanner.
8. potentially confounding medical conditions that impact breathing (e.g.,asthma, congestive heart failure, and emphysema that are not well-controlled), could impact attention to the breath (e.g., chronic pain conditions that are not well-managed), or impact neural functioning (e.g., multiple sclerosis, neurological diseases, brain injury);
9. currently experiencing a mental health condition (e.g., anxiety, depression, panic disorder, post-traumatic stress disorder, attention deficit and hyperactivity disorder) or past severe mental illness such as bipolar disorder, schizophrenia, or severe substance abuse disorder.
10. use of psychotropic medications in the past year
11. current use of medications that potentially can affect the respiratory system or the interoceptive focus in the past week (including narcotics, benzodiazepines); if the research assistant is unclear about a specific medication, the physician on the study (Dr. Rick Hecht) will be asked and will decide;
12. health behaviors that could affect respiration (e.g., DSM-IV diagnosis of substance use disorder, use of major recreational drugs in the past year-heroin, cocaine, etc.);
13. any high-level training in a field that could impact body awareness and is not associated with mind-body practices (e.g., professional athletes or dancers, marathon runners);
14. lack of ability to speak and read English fluently (instructions and questionnaires will be in English only and foreign language translations will have to await future studies);
15. For participants who consent to the fMRI study, exclusion criteria include contra-indications for safety and data quality in the MRI scanner (see MRI screening form): presence of ferromagnetic metal on or in the body, pregnancy, movement disorder which prevents lying still in the scanner, claustrophobia, braces, and corrected vision that is not within +/- 8.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is designed for healthy adults, some of whom have extended meditation practice (at least 5 years), and some who have little or no meditation experience.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Classification accuracy of brain patterns from EMBODY Task | Outcome measure will be assessed once at the baseline fMRI scan to develop the pilot fMRI task.
  The EMBODY Task is a new brain-based measure using functional magnetic resonance imaging (fMRI) to measure meditation skills. The primary outcome measure of the EMBODY Task is whether brain patterns are recognized by pattern classification algorithms for the 5 conditions in the study (attention to breath, body, mind wandering, thoughts, and sounds) above chance levels (20% for 5 conditions, using a one-sample t-test for each condition in the entire sample). Classification accuracy is a standard outcome measure in studies that use brain pattern classification. This will demonstrate that brain patterns associated with internal attention are indeed differentiable by pattern classification methods. These brain patterns will then be used to identify the focus of attention during breath meditation.

SECONDARY OUTCOMES:
Percentage time paying attention to breath during meditation | Outcome measure will be assessed once at the baseline fMRI scan to develop the pilot fMRI task.
  Using EMBODY Task metrics, investigators will calculate how much time people pay attention to their breath during meditation
Percentage time spent mind wandering during meditation | Outcome measure will be assessed once at the baseline fMRI scan to develop the pilot fMRI task.
  Using EMBODY Task metrics, investigators will calculate how much time people were mind wandering during meditation

OTHER OUTCOMES:
Questionnaire measures of attention | Measures will be assessed before the fMRI scan session.
  To validate the EMBODY Task, investigators will administer self-report measures of attention, mindfulness, and body awareness

CONTACTS AND LOCATIONS:
Overall Officials: Helen Y Weng, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators plan to pilot and develop the fMRI EMBODY Task to measure meditation skills, and share any protocols, scripts, and analytic code to administer and analyze the task.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication in the supplementary material
Access Criteria: Available upon publication

REFERENCES:
- [Result] Weng HY, Lewis-Peacock JA, Hecht FM, Uncapher MR, Ziegler DA, Farb NAS, Goldman V, Skinner S, Duncan LG, Chao MT, Gazzaley A. Focus on the Breath: Brain Decoding Reveals Internal States of Attention During Meditation. Front Hum Neurosci. 2020 Aug 28;14:336. doi: 10.3389/fnhum.2020.00336. eCollection 2020. PMID 33005138